CLINICAL TRIAL: NCT03680131
Title: A Randomized, Double-Blind, Vehicle-Controlled, Sample Size Adaptive Design Study to Evaluate the Safety and Efficacy of Topically Applied EB01 Cream in Healthy Adult Volunteers and Adult Subjects with Moderate to Severe Chronic Allergic Contact Dermatitis
Brief Title: Evaluation of EB01 Cream for the Treatment of Chronic Allergic Contact Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Edesa Biotech Inc. (Industry)
Collaborators: JSS Medical Research Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EB01-01-2018
Record Dates: First submitted 2018-09-19; First posted 2018-09-21 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Allergic Contact Dermatitis
MeSH Terms: conditions — Dermatitis, Allergic Contact

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- EB01 Cream Placebo (Active Comparator): EB01 Cream containing 0% EB01 w/w applied BID
  Interventions: Drug: EB01 Cream Placebo
- EB01 Cream 0.2% (Experimental): EB01 Cream containing 0.2% EB01 w/w applied BID
  Interventions: Drug: EB01 Cream 0.2%
- EB01 Cream 1.0% (Experimental): EB01 Cream containing 1.0% EB01 w/w applied BID
  Interventions: Drug: EB01 Cream 1.0%
- EB01 Cream 2.0% (Experimental): EB01 Cream containing 2.0% EB01 w/w applied BID
  Interventions: Drug: EB01 Cream 2.0%

INTERVENTIONS:
Drug: EB01 Cream Placebo — Vehicle Cream containing 0% EB w/w applied BID
  Arms: EB01 Cream Placebo
Drug: EB01 Cream 0.2% — EB01 Cream containing 0.2% EB01 w/w applied BID
  Arms: EB01 Cream 0.2%
Drug: EB01 Cream 1.0% — EB01 Cream containing 1.0% EB01 w/w applied BID
  Arms: EB01 Cream 1.0%
Drug: EB01 Cream 2.0% — EB01 Cream containing 2.0% EB01 w/w applied BID
  Arms: EB01 Cream 2.0%

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of EB01 Cream (0.2%, 1.0%, 2.0%) applied twice per day (BID) for the treatment of moderate to severe chronic allergic contact dermatitis (ACD).

The purpose of the open label extension is to assess the long-term safety, tolerability, and efficacy of EB01 2.0% cream in subjects with moderate to severe chronic allergic contact dermatitis.

ELIGIBILITY:
INCLUSION CRITERIA

All subjects:

1. Men and women ≥ 18 years old, inclusive, at the time of consent.
2. For women of childbearing potential involved in any sexual intercourse that could lead to pregnancy: the subject must agree to use an effective contraceptive method from at least 4 weeks before Day 1 until at least 4 weeks after the last study product application. Effective contraceptive methods include hormonal contraceptives (combined oral contraceptive, patch, vaginal ring, injectable, or implant), intrauterine devices or intrauterine systems, vasectomized partner(s), tubal ligation, or a barrier method of contraception (male condom, female condom, cervical cap, diaphragm, contraceptive sponge) in conjunction with spermicide.

   Note: Subjects must have been on a stable dose of hormonal contraceptives for at least 4 weeks before Day 1.

   Note: The above list of contraceptive methods does not apply to subjects who are abstinent for at least 4 weeks before Day 1 and will continue to be abstinent from penile-vaginal intercourse throughout the study. The reliability of sexual abstinence needs to be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the participant.

   Note: A woman of nonchildbearing potential is as follows:
   1. Woman who has had surgical sterilization (hysterectomy, bilateral oophorectomy, or bilateral salpingectomy);
   2. Woman who has had a cessation of menses for at least 12 months without an alternative medical cause, and a follicle-stimulating hormone (FSH) test confirming nonchildbearing potential (refer to laboratory reference ranges for confirmatory levels).
3. For men involved in any sexual intercourse that could lead to pregnancy, subject must agree to use one of the effective contraceptive methods listed in Inclusion Criterion #2 from Day 1 until at least 4 weeks after the last study product application. If the female partner of a male subject use any of the hormonal contraceptive methods listed above, this contraceptive method must be used by the female partner from at least 4 weeks before Day 1 until at least 4 weeks after the last study product application.
4. Female of childbearing potential has had a negative pregnancy test at screening visit.
5. Subject is willing to participate and is capable of giving informed consent. Note: Consent must be obtained prior to any study-related procedures.
6. Subjects must be willing to comply with all study procedures and must be available for the duration of the study.

HV only:

1. Subject is in good general health, according to the investigator's judgment based on medical history and physical examination/laboratory/ECG/vital signs assessments.

Subjects with allergic contact dermatitis only:

1. Subject has at least 3-month history of allergic contact dermatitis (information obtained from medical chart or subject's physician, or directly from the subject).
2. Subject has moderate to severe chronic allergic contact dermatitis at Day 1, defined by either one of the following:

   * CDSI score ≥ 7
   * CDSI score of severe (3) in ≥ 2 of the 5 assessed symptoms (Fissures, Scaling, Redness, Pruritus, Dryness)
3. Subject has allergic contact dermatitis covering between 0.5% to 10% of the total BSA at Day 1.
4. Subject has an ISGA ≥ 3 at Day 1.
5. The subject has had a positive patch test ("+", "++" or "+++" reaction) to an allergen that is suspected to be involved in the current allergic contact dermatitis in the past 5 years (obtain written documentation of patch test result if possible).

   Alternatively, the Subject agrees to undergo patch testing during the study period (patch testing needs to be completed by Day 36). Guidelines for patch test interpretation are provided in Appendix 2. The measure of the degree of the reaction will be determined on the basis of the reading 2 and 3-4 days post application.
6. Subject agrees to only apply personal care products (i.e. makeup and eyeshadow) that do not contain their allergen(s) on lesions only after applying the IP.
7. Subject agrees not to apply any personal care products on allergic contact dermatitis lesions prior to site visits.

Subjects with allergic contact dermatitis in the Open Label Extension:

1. Subject has completed the main study.

EXCLUSION CRITERIA

All subjects:

1. Subject is a female who is breastfeeding, pregnant, or who is planning to become pregnant during the study.
2. Current or recurrent disease, other than allergic contact dermatitis (applicable to subject with allergic contact dermatitis only), that could affect the action, absorption, or disposition of the study drug, or clinical or laboratory assessments.
3. Subject has a history of skin disease or presence of skin condition, other than allergic contact dermatitis (applicable to subject with allergic contact dermatitis only) that, in the opinion of the investigator, would interfere with the study assessments.
4. Subject is known to have immune deficiency or is immunocompromised.
5. Subject has a history of cancer or lymphoproliferative disease within 5 years prior to Day 1. Subjects with successfully treated non-metastatic cutaneous squamous cell or basal cell carcinoma and/or localized carcinoma in situ of the cervix are not to be excluded.
6. Subject had a major surgery within 8 weeks prior to Day 1 or has a major surgery planned during the study.
7. Subject has any clinically significant medical condition that would, in the opinion of the investigator, put the subject at undue risk or interfere with interpretation of study results.
8. Subject has a known history of chronic infectious disease (e.g., hepatitis B, hepatitis C, or infection with human immunodeficiency virus).
9. Subject has used systemic treatments (other than biologics) that could affect allergic contact dermatitis (applicable to subjects with allergic contact dermatitis only) or is known to cause cutaneous irritation or sensitization reactions less than 2 weeks prior to Day 1 (e.g., oral/injectable corticosteroids, retinoids, calcineurin inhibitors, methotrexate, cyclosporine, hydroxycarbamide [hydroxyurea], azathioprine) Note: Intranasal corticosteroids and inhaled corticosteroids for stable medical conditions are allowed. Eye drops containing corticosteroids are allowed.
10. Use of any prescription or over-the-counter (OTC) medication that, in the opinion of the Principal Investigator, could affect (improve or worsen) the allergic contact dermatitis condition or is known to cause cutaneous irritation or sensitization reactions.
11. Subject has received any marketed or investigational biological agent within 12 weeks or 5 half-lives (whichever is longer) prior to Day 1.
12. Subject is currently receiving a nonbiological investigational product or device or has received one within 2 weeks prior to Day 1.
13. Subject has received any UV-B phototherapy (including tanning beds) or excimer laser within 2 weeks prior to Day 1.
14. Subject had excessive sun exposure, is planning a trip to a sunny climate, or has used tanning booths within 2 weeks prior to Day 1 or is not willing to minimize natural and artificial sunlight exposure during the study. Use of sunscreen products and protective apparel are recommended when exposure cannot be avoided. If sunscreen is applied to ACD lesions, it should be applied after the IP.
15. Subject has a known hypersensitivity to EB01 or its excipients.
16. Subject has uncontrolled diabetes.
17. Subject has a known history of clinically significant drug or alcohol abuse in the last year prior to Day 1.

HV only:

1. Subject has history of recurrent chronic or presence of allergic contact dermatitis.
2. Subject has used any medicated topical product on the face within 2 weeks prior to Day 1.

Subjects with allergic contact dermatitis only:

1. Subjects with active atopic dermatitis lesions overlapping with allergic contact dermatitis lesions at Day 1.
2. Subject has clinically infected allergic contact dermatitis lesions (bacterial, viral, or fungal).
3. Subject has allergic contact dermatitis on lips or mucous membranes only.
4. Subject has used dupilumab within 12 weeks prior to Day 1.
5. Subject has used doxepin within 1 week prior to Day 1.
6. Subject has used hydroxyzine or diphenhydramine within 1 week prior to Day 1.
7. Subject has used topical products containing urea within 1 week prior to Day 1.
8. Subject has used systemic antibiotics within 2 weeks or topical antibiotics on lesions of allergic contact dermatitis within 1 week prior to Day 1.
9. Subject has used any topical medicated treatment for allergic contact dermatitis within 1 week prior to Day 1, including, but not limited to, topical corticosteroids, crisaborole and any other topical phosphodiesterase-4 inhibitor, calcineurin inhibitors, tars, bleach, antimicrobials and medical devices.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 211 (Actual)
Dates: Start 2019-10-15 (Actual); Primary Completion 2022-09-21 (Actual); Study Completion 2023-01-17 (Actual)

PRIMARY OUTCOMES:
Mean percent change from baseline in the Contact Dermatitis Severity Index (CDSI) | Day 29

SECONDARY OUTCOMES:
Mean percent change from baseline in CDSI | Days 15, 59, 89, and 119
Proportion of subjects achieving at least a 2-grade reduction from baseline to clear (0) or almost clear (1) in Investigator's Static Global Assessment (ISGA) | Days 15, 29, 59, 89, and 119
Mean percent change from baseline in Body Surface Area (BSA) affected with chronic allergic contact dermatitis | Days 15, 29, 59, 89, and 119
Change from baseline in Dermatology Life Quality Index (DLQI) | Days 15, 29, 59, 89, and 119
Proportion of patients achieving at least a 2-point reduction from peak pruritis Numerical Rating Scale (NRS) score from Baseline | Days 15, 29, 59, 89, and 119
Proportion of patients achieving at least a 4-point reduction from peak pruritis Numerical Rating Scale (NRS) score from Baseline | Days 15, 29, 59, 89, and 119

OTHER OUTCOMES:
Treatment-emergent adverse events (TEAEs) | To Day 36, and for open-label extension to Day 119
  Number of events
Safety and tolerability assessments | To Day 36, and for open-label extension to Day 119
  Changes in vital signs, physical examinations, ECG, safety laboratory tests, and local tolerability assessment. Tolerability will be assessed using a numerical rating scale from 0 to 10, and will evaluate skin burning, stinging and pruritus during treatment

CONTACTS AND LOCATIONS:
Locations (15):
- United States (14):
  - Ark Clinical Research, Long Beach, California
  - Foxhall Dermatology, Washington D.C., District of Columbia
  - Gold Coast Dermatology, Delray Beach, Florida
  - Miami Dade Medical Research Institute, LLC, Miami, Florida
  - The Dermatology Centre of Indiana, Plainfield, Indiana
  - Forefront Dermatology, Louisville, Kentucky
  - The Dermatology Clinic, Baton Rouge, Louisiana
  - Oakland Hills Dermatology P.C., Auburn Hills, Michigan
  - Associated Skin Care Specialists, Fridley, Minnesota
  - JUVA Skin & Laser Center, New York, New York
  - UNC Dermatology and Skin Cancer Center, Chapel Hill, North Carolina
  - Bexly Dermatology, Bexley, Ohio
  - Apex Clinical Research Center, LLC, Mayfield Heights, Ohio
  - West Virginia Research Institute, Morgantown, West Virginia
- Lynderm Research Inc., Markham, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No